CLINICAL TRIAL: NCT00898521
Title: Feasibility Study: Enzymatic Debridement in Patients With Partial Thickness Burns (Children & Adults)- Protocol MW2008-09-03
Brief Title: Feasibility Study: Enzymatic Debridement in Patients With Partial Thickness Burns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MW2008-09-03
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2011-04

CONDITIONS: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DGD (Experimental)
  Interventions: Drug: DGD

INTERVENTIONS:
Drug: DGD — DGD is a mixture of lyophilized enzymes derived from purified Bromelain from pineapple stem.
  Two grams or 5 grams of Debrase powder are dissolved in 20 grams or 50 grams of Gel Vehicle to obtain DGD. DGD is applied to the burn wound at a dose of 2g Debrase/20g Gel per 100 cm2 of skin or 5g Debrase/50g Gel per 250 cm2 for a duration of four hours. In an average human adult, 100 cm2 represents approximately 1% of Total Body Surface Area (TBSA).
  Please note that for individuals of exceptional size (e.g. children), it is important to calculate the dosage based on the 100 cm2 measurement.
  The Debrase powder and the Gel Vehicle are to be mixed at the patient bedside for a maximum of 15 min prior to use.
  DGD should not be applied to more than 15% TBSA in one session. If the wound area to be treated is more than 15% TBSA, DGD should be applied in two or more separate sessions.
  DGD should not be applied more than twice to the same burn wound area.

SUMMARY:
Burns represent one of the most severe and dreaded traumas. Burned and traumatized tissue is known as eschar. The dead eschar, if not removed, often becomes heavily contaminated and is the source of local and/or systemic infection or sepsis. The local inflammation and infection destroy healthy surrounding tissues and extends the original damage. In order to prevent these complications, and in order to minimize the risk of infection, it is imperative to evaluate the burn and remove all of the offending eschar at the earliest possible opportunity. This removal of dead tissue is termed "debridement".

The most direct debridement method for eschar removal is surgery. Traditional, conservative non-surgical debridement is a lengthy process which often involves many complications.

The objectives of this study are as follows:

1. To evaluate the safety and efficacy (exploratory) of DGD in hospitalized patients with Partial Thickness (mid and deep dermal) thermal burns of 4-30% total body surface area (TBSA), but with total burn wounds of no more than 30% TBSA. Measures have already been taken in previous studies involving deeper wounds to control safety parameters (such as pain, fever and infection). Nevertheless, as part of the effort to expand the burn population in the future phase 3 study to the more superficial wound group, it is important to first explore these parameters in a small group involving this burn population.
2. To explore DGD absorption as measured by Pharmacokinetic testing.

DETAILED DESCRIPTION:
on-going recruitment, children and adults

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 2 years and 55 years of age,
2. Thermal burns caused by fire/flame, scalds or contact,
3. Burn composition must be as follows:

   1. Partial Thickness (mid & deep dermal) burn wounds ≥ 4% and ≤ 30% Total Body Surface Area (TBSA),
   2. Full thickness burns ≤ 5%,
4. All the partial and full thickness burn wounds must receive study treatment except facial, genital or perineal burns (Exclusion Criteria #5 and #6 below),
5. Total burn wounds ≤ 30% TBSA,
6. Hospital admission within 24 hours of the burn injury. Patients transferred from another hospital/clinic may be enrolled if the primary admission was within 24 hours of the burn injury and admission to the burn unit participating in the study was within 48 hours of the burn injury,
7. Signed written informed consent.

Exclusion Criteria:

1. More than 5% TBSA full thickness burns,
2. Patient having only full thickness burns,
3. Other severe cutaneous trauma at the same sites as the burns (i.e. considerable blunt, avulsion or deep abrasion), or previous burn(s) at the same treatment site(s),
4. One or more burn wounds that do not meet study criteria,
5. Deep partial thickness and/or full thickness facial burn wounds >0.5% TBSA; study treatment of facial burns is not allowed,
6. Study treatment of perineal and/or genital burns is not allowed; A patient with these wounds may be enrolled but the wounds may not be designated as target wounds,
7. Patient with circumferential anterior/posterior trunk fire/flame burns, >15% TBSA Circumferential is defined as encircling ≥ 80% of the trunk circumference),
8. A. The following pre enrolment dressings: a. Flammacerium, b. Silver Nitrate AgNO3), B. Pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by pseudoeschar (e.g. pseudoeschar as a result of SSD treatment);
9. Pre-enrolment escharotomy,
10. Heavily contaminated burns or pre-existing infections (Adults: WBC ≥ 20.0 X 103 cells/µL; Children aged 4-18: WBC ≥ 25.0 X 103 cells/µL)),11.Signs that may indicate smoke inhalation (e.g. clinical signs, etiology of injury, venue of injury, etc.),
11. Children with Hb < 10 gm/dl at Screening/Pre treatment
12. Prisoners,
13. Pregnant women (positive pregnancy test) or nursing mothers,
14. Poorly controlled diabetes mellitus (HbA1c>9%),
15. Cardio-pulmonary disease (MI within 4 weeks prior to injury, pulmonary hypertension, COPD or pre-existing oxygen-dependent pulmonary diseases),
16. Pre-existing diseases which interfere with circulation (PVD, edema, lymphedema, surgery to the regional lymph nodes, obesity, varicose veins),
17. Immediate life threatening conditions (such as immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder, cardiovascular, liver or neoplastic disease),
18. Chronic systemic steroid intake,
19. History of allergy and/or known sensitivity to pineapples or papain,
20. Current suicide attempt,
21. Participation in another investigational drug trial,
22. Current alcohol or drug abuse,

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12-20 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is safety as measured by: 1. Systemic an local adverse events, 2. Changes in vital signs and laboratory tests, 3. Time to wound closure. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Lior Rosenberg, MD, Study Chair — MediWound Ltd
Locations (2):
- Lok Nayak hospital, New Delhi, India
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Rosenberg L, Lapid O, Bogdanov-Berezovsky A, Glesinger R, Krieger Y, Silberstein E, Sagi A, Judkins K, Singer AJ. Safety and efficacy of a proteolytic enzyme for enzymatic burn debridement: a preliminary report. Burns. 2004 Dec;30(8):843-50. doi: 10.1016/j.burns.2004.04.010. PMID 15555800